CLINICAL TRIAL: NCT02279108
Title: Comparative, Prospective, Randomized Study Assessing The Interest of Indocyanine Green Fluorescence Imaging With Radioisotope Method For Sentinel Lymph Node Biopsy in Patients With Breast Cancer
Brief Title: Study Assessing The Interest of Indocyanine Green Fluorescence Imaging With Radioisotope Method For Sentinel Lymph Node Biopsy in Patients With Breast Cancer
Acronym: FLUOTECH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1408153; 2014-004005-32 (EudraCT Number)
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2017-09

CONDITIONS: Breast Neoplasms
Keywords: sentinel lymph node; indocyanine green; fluorescence method; radioisotope conventional method; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green; Isotopes; Technetium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- double detection Indocyanine + isotope (Experimental): intradermal injection of 2.5 milligrams of indocyanine green and 20 MBq of technetium 99 before breast surgery
  Interventions: Drug: indocyanine green; Drug: isotope
- isotope detection alone (Active Comparator): intradermal injection of 20 MBq of technetium 99 before breast surgery
  Interventions: Drug: isotope

INTERVENTIONS:
Drug: indocyanine green — One injection, 2.5 milligrams per patient, intradermal use
  Arms: double detection Indocyanine + isotope
Drug: isotope — One injection, 20 MBq techntium99, intradermal use
  Other Names: technetium

SUMMARY:
The sentinel node has a fundamental role in the management of early breast cancer.

Currently, the double detection of blue and radioisotope is recommended. A radioactive material requires the presence of a nuclear medicine department and the approval of health authorities. In many centers, this technique is not available. The use of blue is easier to implement technique. However, allergic reactions and prolonged breast tattoo led many teams to stop the practice.

So in common practice, many center use a single method. However, with a single detection, the risk of false negatives and the identification failure rate increased to a significant extent and the number of sentinel lymph node detected and removed is not enough.

Under these conditions, find another method of detection seems crucial. According to the literature, the fluorescence method (ICG) is a technique that seems safe and reliable.

The investigators therefore propose a prospective, randomized study to investigate the interest of fluorescence associated with the isotopic method.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved infiltrating breast cancer (ductal, lobular carcinoma…) or a carcinoma in-situ with an elevated risk of micro-invasion. (High grade with necrosis, radiologically evaluated size more than 40mm, or immediate mastectomy…)
* Unifocal or multifocal but in same quarter
* Size < 5cm clinically palpable or not
* Clinically or ultrasound axillary N0
* Isotopic sentinel node detection
* Adult patient
* Signed informed consent by patient or legally responsable authority
* Patient registered to a social security system
* No surgical contra-indication

Exclusion Criteria:

* Mammary carcinoma recurrence
* Previous same side mammary reduction
* Previous lumpectomy
* Contra-indication to surgery
* Pregnant or breast feeding patient
* Denial of participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Céline CHAULEUR, PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
Started | 50 | 50
Completed | 50 | 49
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (12.0) | 60.2 (12.5) | 61.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 99
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
height, continuous [Mean (Standard Deviation); unit: cm] | 161.1 (5.4) | 160.4 (6.1) | 160.8 (5.7)
weight, continuous [Mean (Standard Deviation); unit: kg] | 69.6 (13) | 65.0 (11.1) | 67.3 (12.3)
age of first menstruation, continuous [Mean (Standard Deviation); unit: years] — Population: data not find
  years
    number analyzed (Participants) | 47 | 40 | 87
    (all) | 12.8 (1.5) | 12.8 (1.4) | 12.8 (1.5)
menopause [Count of Participants; unit: Participants] — Population: Data not found
  Participants
    number analyzed (Participants) | 50 | 48 | 98
    (all) | 34 | 30 | 64
tumor size [Median (Inter-Quartile Range); unit: mm] — Population: data not found
  mm
    number analyzed (Participants) | 49 | 48 | 97
    (all) | 15 [10 to 25] | 15 [11 to 22.5] | 15 [10 to 23.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Less Than Two Lymph Nodes Detected
Description: Number of patients with less than two lymph nodes detected by indocyanine (ICG) + isotope versus isotope detection alone
Time Frame: peroperative
Measure: Count of Participants; unit: Participants
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
Number analyzed (Participants) | 50 | 49
Participants | 22 | 20

2. Secondary Outcome: Number of Lymph Nodes ICG Positive and Tc Positive
Description: Number of lymph nodes Indocyanine green (ICG) positive and Tc (Technetium)positive
Time Frame: Peroperative
Measure: Number; unit: lymph nodes
Units Other Than Participants: lymph nodes
Arm/Group | Double Detection Indocyanine + Isotope
Number analyzed (Participants) | 50
Number analyzed (lymph nodes) | 108
lymph nodes | 85

3. Secondary Outcome: Number of Lymph Nodes ICG Positive and Tc Negative
Description: Number of lymph nodes Indocyanine green (ICG) positive and Tc (Technetium) negative
Time Frame: Peroperative
Measure: Number; unit: lymph nodes
Units Other Than Participants: Lymph nodes
Arm/Group | Double Detection Indocyanine + Isotope
Number analyzed (Participants) | 50
Number analyzed (Lymph nodes) | 108
lymph nodes | 15

4. Secondary Outcome: Number of Lymph Nodes ICG Negative and Tc Positive
Description: Number of lymph nodes Indocyanine green (ICG) negative and Tc (Technetium) positive
Time Frame: Peroperative
Measure: Number; unit: lymph nodes
Units Other Than Participants: lymph nodes
Arm/Group | Double Detection Indocyanine + Isotope
Number analyzed (Participants) | 50
Number analyzed (lymph nodes) | 108
lymph nodes | 7

5. Secondary Outcome: Comparison Between Groups of the Time of the Surgery
Description: time from incision to wound closure
Time Frame: Peroperative
Measure: Median (Inter-Quartile Range); unit: minuts
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
Number analyzed (Participants) | 50 | 49
minuts | 92.5 [72 to 122] | 76 [59 to 98]

6. Secondary Outcome: Comparison Between Groups of Anesthesia Time
Description: time from the injection of anesthesic to the waking
Time Frame: Peroperative
Measure: Median (Full Range); unit: minutes
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
Number analyzed (Participants) | 49 | 48
minutes | 171 [95 to 301] | 152 [85 to 365]

7. Secondary Outcome: Time From Injection of One Dose ICG Injection to Incision Time
Description: time from injection of one dose ICG injection to incision time
Time Frame: Peroperative
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Double Detection Indocyanine + Isotope
Number analyzed (Participants) | 50
minutes | 17.5 [13 to 24]

8. Secondary Outcome: Comparison Between Groups of Time Surgery Node
Description: time from incision time to the last node surgery
Time Frame: Peroperative
Measure: Median (Inter-Quartile Range); unit: minuts
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
Number analyzed (Participants) | 49 | 48
minuts | 171 [142 to 200] | 162.3 [125 to 194]

9. Secondary Outcome: Number of Patients With ICG Allergy
Description: allergy is : redness, edema, itching, larynges edema and/or allergic shock
Time Frame: peroperative
Measure: Count of Participants; unit: Participants
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
Number analyzed (Participants) | 50 | 49
Participants | 0 | 0

10. Secondary Outcome: Number of Patients With ICG Allergy
Description: allergy is : redness, edema, itching, larynges edema and/or allergic shock
Time Frame: 1 hour after the end of the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
Number analyzed (Participants) | 50 | 49
Participants | 0 | 0

11. Secondary Outcome: Number of Patients With ICG Allergy
Description: allergy is : redness, edema, itching, larynges edema and/or allergic shock
Time Frame: Month 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
Number analyzed (Participants) | 50 | 49
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Double Detection Indocyanine + Isotope | Isotope Detection Alone
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 16/50 | 13/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Detection Indocyanine + Isotope (N=50) | Isotope Detection Alone (N=49)
hematoma (Surgical and medical procedures) | 5 (5) | 7 (7)
lymphocele (Blood and lymphatic system disorders) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No